CLINICAL TRIAL: NCT05398861
Title: A Single-arm, Prospective, Open-label Phase II Clinical Study of Utidelone Combined With Bevacizumab in the Treatment of ≥ 2 Lines of HER-2 Negative Advanced Breast Cancer
Brief Title: Utidelone Combined With Bevacizumab in the Treatment of ≥ 2 Lines of HER-2 Negative Advanced Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Collaborators: Qilu Pharmaceutical Co., Ltd. (Industry); Beijing Biostar Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HNCH-MBC11
Record Dates: First submitted 2022-05-22; First posted 2022-06-01 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-04

CONDITIONS: HER-2 Negative Breast Cancer
MeSH Terms: interventions — Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HER-2 Negative Advanced Breast Cancer (Experimental): Utidelone Combined with Bevacizumab
  Interventions: Drug: Utidelone Combined with Bevacizumab

INTERVENTIONS:
Drug: Utidelone Combined with Bevacizumab — Utidelone： 30 mg/m2/day, IV transfusing over 90 min. on day 1-day 5 of each 21 day cycle Bevacizumab：10mg/kg (IV), on day 1 of each 21 days.
  Other Names: UTD1

SUMMARY:
This study is a prospective, single-arm, open-label phase II study to evaluate the efficacy and safety of the combination of Utidelone and bevacizumab regimen in patients with ≥ 2 lines of HER-2 negative advanced breast cancer.

DETAILED DESCRIPTION:
Patients included were patients with ≥ 2 lines of HER2-negative advanced breast cancer who had previously failed taxanes and/or anthracyclines, or patients with hormone receptor-positive HER2-negative advanced breast cancer who had progressed after at least 1 line of prior endocrine therapy.

This study used a Simon two-stage design. 71 subjects will be enrolled using the optimal design.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form;
2. Women aged 18-70 years;
3. The number of treatment lines for patients ≥ 2 lines；
4. Histologically or cytologically confirmed HER2-negative locally advanced or metastatic breast cancer:
5. Patients with HER2-negative breast cancer who have failed previous treatment with taxanes and/or anthracyclines, or patients with hormone receptor-positive HER2-negative advanced breast cancer who have progressed after at least one line of previous endocrine drug therapy;
6. Eastern Cooperative Oncology Group (ECOG) score [0-2] points，Life expectancy of not less than 3 months；
7. At least one evaluable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST1.1)；
8. Adequate hematological, hepatic and renal function；
9. Patients must have recovered to ≤ Grade 1 (CTCAE v5.0) from all toxicities related to prior anticancer therapy；
10. Women of childbearing age must agree to use highly effective methods of contraception during the study and within 6 months after administration of the study drug; Subjects must be non-lactating and have a negative serum or urine pregnancy test within 7 days prior to study enrollment

Exclusion Criteria:

1. Patients who have progressed on prior bevacizumab；
2. Patients who have previously used Utidelone, and the interval is less than 6 months from the end of medication；
3. Less than 3 weeks after radiotherapy or chemotherapy; less than 1 week after endocrine therapy；
4. Concomitant diseases/medical history； （1）Clinically significant hemoptysis (with daily hemoptysis of more than 50 ml) within 3 months before enrollment; or clinically significant bleeding symptoms or definite bleeding tendency, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, fecal occult blood or greater at baseline, or suffering from vasculitis； （2）Patients with arteriovenous thrombotic events within 6 months before enrollment, such as cerebrovascular accident (including transient ischemic attack), deep venous thrombosis (except resolved venous thrombosis caused by previous chemotherapy, which has been judged by the investigator) and pulmonary embolism； （3）Hypertension not adequately controlled with antihypertensive therapy (systolic blood pressure > 140 mmHg or diastolic blood pressure > 90 mmHg); Randomization occurs within 6 months as follows: myocardial infarction, severe/unstable angina, NYHA Class 2 or greater, clinically significant supraventricular or ventricular arrhythmia, and symptomatic congestive heart failure （4）Interstitial lung disease, pneumonitis, or uncontrollable systemic disease (e.g., diabetes, pulmonary fibrosis, acute pneumonitis, etc.； （5）Renal insufficiency: urine routine showed urine protein ≥ + +, or 24 h urine protein ≥ 1.0g was confirmed； （6）History of attenuated live vaccine within 28 days before the first dose of study drug or anticipated vaccination with live attenuated vaccines during the study （7）Human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS); active hepatitis (hepatitis B, defined as HBV-DNA ≥ 500 IU/ml; hepatitis C, defined as HCV-RNA above the lower limit of detection of the analytical method) or co-infection with hepatitis B and C； （8）Presence of severe infection within 4 weeks before administration, including but not limited to bacteremia requiring hospitalization, severe pneumonia, etc. Active infection with CTCAE 5.0 ≥ grade 2 requiring systemic antibiotic therapy within 2 weeks before the first dose, or unexplained fever > 38.5 ° C during the screening period/before the first dose (fever due to tumor causes may be included if judged by the investigator); evidence of active tuberculosis infection within 1 year before dosing.
5. Any other malignancy diagnosed within 3 years before study entry；
6. Major surgery within 28 days and minor surgery within 14 days before enrollment；
7. Patients who have previously received or are ready to receive allogeneic bone marrow transplantation or solid organ transplantation；
8. Peripheral neuropathy ≥ grade 2; active brain metastases, carcinomatous meningitis, spinal cord compression, or brain or leptomeningeal disease found by CT or MRI at screening (patients with brain metastases who have completed treatment on 14 days before enrollment and have stable symptoms, however, it needs to be confirmed as no cerebral hemorrhage symptoms by brain MRI, CT or venography evaluation);
9. Female patients who are pregnant, lactating, or plan to become pregnant during the study;
10. Patients who have other serious physical or mental illness or abnormal laboratory findings that may increase the risk of study participation, or interfere with study results, and are not suitable for this study in the opinion of the investigator;

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | up to 2 years
  Percentage of patients with a best investigator-assessed response of CR or PR from enrollment until disease progression as assessed by RECIST 1.1 compared with the total number of evaluable patients.

SECONDARY OUTCOMES:
Progression free survival (PFS) | up to 2 years
  PFS is defined as the duration of time from first study treatment to disease progression or death from any cause as documented by the investigator
Overall survival (OS) | up to 3 years
  OS is defined as the duration of time from first study treatment until death from any cause.

IPD SHARING:
Plan to Share IPD: No
Due to the small sample size in this trial, Individual Patient Data cannot be adequately anonymized and there is a reasonable likelihood that individual participants could be re-identified. For this reason, data from this trial cannot be shared.